CLINICAL TRIAL: NCT05127863
Title: Efficacy of a Pragmatic Intervention to Improve Adaptation to Context and Interlocutor
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is completed
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRAGMA-INTERV
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Autism Spectrum Disorder; Developmental Language Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Language Development Disorders

STUDY DESIGN:
Intervention Model Description: multiple single case study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2 to 5 ASD or TDL patients (Experimental): 2 to 5 ASD or TDL patients, 8 to 14 years old, with no intellectual disability.
  Interventions: Behavioral: social communication intervention (pragmatic)

INTERVENTIONS:
Behavioral: social communication intervention (pragmatic) — 10 sessions of group intervention in order to improve pragmatic/social communication. one session of one hour per week. Activities will included role play, conversations, etc.

SUMMARY:
Patients with Developmental Language Disorder (DLD) or Autism Spectrum Disorder (ASD) have communicational difficulties to adapt their language to context and to interlocutors. These difficulties have long term impacts on education and social life of these patients. Speech language therapists (SLT) helps child and teenagers with pragmatic and communicational disorders. Nevertheless, few research evaluated the efficacy of such interventions.

In the present research, the students will do a literature review to identify efficacy intervention's strategies of pragmatic disorders. Then, 2 to 5 patients, aged from 8 to 14 years old, with ASD or DLD and pragmatic disorders, and who haven't intellectual disorder will be recruited. They will come to the faculty of psychology of UCLouvain before the beginning of the intervention. In this pretest session, parents will answer questionnaires et children will have tests in order to evaluate their pragmatic abilities (during 30 minutes), like conversations, role plays, communication referential tasks, etc. This evaluation will be video recorded to code pragmatic abilities. Then, a group intervention of ten sessions will be proposed (1 session per week, 10 weeks). Activities will include role plays, conversations, etc. At the end of the intervention period, a post test session, like the pretest session, will be proposed to evaluate intervention efficacy.

The design is multiple study cases. This is the best design to control efficacy of these kind of interventions considering the inter-individual variability of DLD and ASD patients. This study is original since few research evaluated the efficiency of pragmatic intervention. Some studies demonstrated the efficacy of pragmatic intervention in DLD and ASD patients but theses researches were conducted in English-speaking countries. Furthermore, the present research will propose a group intervention, which weren't proposed in the literature to our knowledge (individual intervention). If the group intervention is efficacy, the cost-benefice ratio would be interested.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic of ASD or DLD
* pragmatic difficulties

Exclusion Criteria:

* intellectual deficiency

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
social communication abilities (according parents) | through study completion, an average of 6 months
  questionnaire (Children Communication Checklist) - pragmatic scale Maximum 162 (good performance), minimum 86 (bad performance)
social communication abilities (evaluated by clinician) | through study completion, an average of 6 months
  social communication task, conversations

CONTACTS AND LOCATIONS:
Locations (1):
- UCLouvain - faculty of psychology, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No